CLINICAL TRIAL: NCT02784262
Title: Botulinum Toxin Type A Block of the Sphenopalatine Ganglion in Chronic Rhinosinusitis With Nasal Polyposis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 011015-01; 2015-004377-33 (EudraCT Number)
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Chronic Disease; Nasal Polyposis; Rhinitis
Keywords: Botulinum Toxin Type A; Block; Sphenopalatine Ganglion
MeSH Terms: conditions — Chronic Disease; Nasal Polyps; Rhinitis; Bites and Stings | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- botox injection (Experimental): * Preoperative medication: Paracetamol 1,5g oral, diclofenac 50mg (evt ibuprofen 600mg) oral and/or diazepam 5-10 mg oral.
  * Skin and tissue inside the projected injection canal will be infiltrated with 5-10ml Marcain-Adrenalin (5mg/ml + 5microg/ml) for local anaesthesia.
  * Localization will be confirmed with help of navigation before the medication will be given. Intravascular injection will be prevented by control of aspiration.
  Interventions: Drug: botox injection Multiguide

INTERVENTIONS:
Drug: botox injection Multiguide — botox injection under CT/MR navigation and with the navigation tool MultiGuide
  Other Names: Botulinum toxin type A

SUMMARY:
Chronic rhinosinusitis (CRS) with nasal polyps is a particularly challenging form of chronic rhinosinusitis in several ways. Patients have significantly more severe symptom burden and worse quality of life than patients with chronic rhinosinusitis without nasal polyps. Many patients return to the health care providers with persistent symptoms after repeated medical and surgical treatment. Patients have usually tried several different types of treatments, ranging from less invasive procedures to extensive surgical treatment. The surgical treatment is often repeated several times. The most common surgical treatment is functional endoscopic sinus surgery, another established procedure is Vidian neurectomy.

The main object of this pilot study is to investigate the safety of onabotulinumtoxin A towards the sphenopalatine ganglion (SPG) in CRS patients with nasal polyps. Efficacy data will also be collected to provide indication on whether future placebo-controlled studies should be performed.

Onabotulinumtoxin A inhibits the secretion of acetylcholine, blocking the parasympathetic reflex cascade in the SPG. As a result, the investigators expect less mucosal swelling, secretion and nasal polyps. The duration of such a blockade is believed to last for 3-9 months and will not lead to damage of the nerve.

This study opens up for improved treatment with less complications.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* chronic rhinosinusitis with nose polyps (CRSwNP) according to European position paper on rhinosinusitis and nasal polyps (EPOS) criteria
* no satisfactory effect of medicinal or surgical treatment

Exclusion Criteria:

* systemic or local disease or condition that may result in a higher risk for complications
* psychiatric disorder that is indicates against the treatment
* pregnancy, breastfeeding, fertile female not using contraception
* abuse of drugs, narcotics or alcohol
* hypersensitivity against marcain, lidocain, xylocain, or adrenalin, and similar drugs
* anatomical conditions that hinder injection
* known sensitivity for botulinum toxin type A or for adjuvant substances
* treatment with drugs that interact with botulinum toxin type A:
* suspicion of polyps caused by an allergy
* suspicion of Samters triade

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
adverse events | from day 1 to 7 post surgery
  Registration of all adverse events sorted by probable relation to botox or surgery. Data collected from symptom diary, in addition to an open question at consultation and put into the Case Report Form (CRF) by physician or nurse.

SECONDARY OUTCOMES:
change in symptom index on a visual analog scale nasal obstruction/running nose | 3 months
change in sinonasal quality of life assessed with the sino-nasal outcome test 22 (SNOT-22) | 3 months
change in nose-sinus related quality of life assessed with a visual analog scale (VAS) | 3 months
change in the geometrics of the nose assessed by acoustic rhinometry | 3 months
change in air flow in the nose measured by peak nasal inspiratory flow (PNIF) | 3 months
change in polyp mass assessed by magnetic resonance imaging (MRI) | 3 months
change in polyp mass assessed by computer tomography (CT) | 3 months
change in quality of life expressed by Patients' Global Impression of Change (PGIC) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lars Jacob Stovner, md prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Jamtoy KA, Tronvik E, Bratbak DF, Crespi J, Stovner LJ, Aschehoug I, Thorstensen WM. OnabotulinumtoxinA injection towards the SPG for treating symptoms of refractory chronic rhinosinusitis with nasal polyposis: a pilot study. Acta Otolaryngol. 2021 Oct;141(10):934-940. doi: 10.1080/00016489.2021.1982146. Epub 2021 Oct 11. PMID 34633904